CLINICAL TRIAL: NCT04677504
Title: A Phase II, Randomized, Double-Blind Placebo-Controlled Study of Atezolizumab With or Without Bevacizumab in Combination With Cisplatin Plus Gemcitabine in Patients With Untreated, Advanced Biliary Tract Cancer
Brief Title: A Study of Atezolizumab With or Without Bevacizumab in Combination With Cisplatin Plus Gemcitabine in Patients With Untreated, Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO42661
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — atezolizumab; Bevacizumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Atezo+Bev+CisGem, followed by Atezo+Bev (Experimental): Participants will receive atezolizumab intravenously on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, and clinical status. Participants will receive bevacizumab intravenously on Day 1 of each 21-day cycle. Participants will receive cisplatin intravenously followed by gemcitabine on Days 1 and 8 of each 21-day cycle for Cycles 1-8.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Cisplatin; Drug: Gemcitabine
- Arm B: Atezo+PBO+CisGem, followed by Atezo+PBO (Active Comparator): Participants will receive atezolizumab intravenously on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, and clinical status. Participants will receive placebo matching bevacizumab intravenously on Day 1 of each 21-day cycle. Participants will receive cisplatin intravenously followed by gemcitabine on Days 1 and 8 of each 21-day cycle for Cycles 1-8.
  Interventions: Drug: Atezolizumab; Other: Placebo; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered intravenously at a fixed dose of 1200 mg on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 mg/kg intravenously on Day 1 of each 21-day cycle after atezolizumab.
  Other Names: Avastin
  Arms: Arm A: Atezo+Bev+CisGem, followed by Atezo+Bev
Other: Placebo — Placebo matching bevacizumab will be administered intravenously on Day 1 of each 21-day cycle after atezolizumab.
  Arms: Arm B: Atezo+PBO+CisGem, followed by Atezo+PBO
Drug: Cisplatin — Cisplatin will be administered intravenously at a dose of 25 mg/m^2 on Days 1 and 8 of each 21-day cycle for Cycles 1-8.
Drug: Gemcitabine — Gemcitabine will be administered intravenously at a dose of 1000 mg/m^2 on Days 1 and 8 of each 21-day cycle for Cycles 1-8.

SUMMARY:
This study will evaluate the efficacy and safety of atezolizumab with bevacizumab in combination with cisplatin and gemcitabine(CisGem), compared with atezolizumab in combination with CisGem, in participants with advanced biliary tract cancer (BTC) who have not received prior systemic therapy. Treatment will consist of a chemotherapy combination phase followed by a cancer immunotherapy (CIT)/placebo phase.

ELIGIBILITY:
Inclusion Criteria:

* Considered to be eligible to receive platinum-based chemotherapy, in the investigator's judgment
* Documentation of recurrent/metastatic or locally advanced unresectable disease based on computed tomography (CT) or magnetic resonance imaging (MRI) scans
* Histologically or cytologically confirmed diagnosis of iCCA, eCCA, or GBC
* No prior systemic therapy for advanced BTC
* At least one measurable untreated lesion (per RECIST v1.1)
* Adequate biliary drainage with no evidence of ongoing infection
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Life expectancy of > 3 months
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Recurrent disease <=6 months after curative surgery or <= 6 months after the completion of adjuvant therapy
* Prior local regional therapy such as radioembolization
* Combined or mixed hepatocellular/cholangiocarcinoma
* Clinically significant hepatic encephalopathy within the 12 months prior to Day 1 of Cycle 1
* National Cancer Institute Common Terminoogy Criteria for Adverse Events Grade >= 2 peripheral neuropathy
* Prior bleeding event due to untreated or incompletely treated esophageal and/or gastric varices within 6 months prior to Day 1 of Cycle 1
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of atezolizumab or within 6 months after the final dose of bevacizumab, cisplatin or gemcitabine
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* History of malignancy other than BTC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Symptomatic, untreated, or actively progressing CNS metastases
* For patients with lung metastases, if one of the following criteria applies: Large, centrally located pulmonary metastases; Clear tumor infiltration into the thoracic great vessels seen on imaging; Clear cavitation of pulmonary lesions seen on imaging
* Active tuberculosis
* Co-infection with HBV and HCV
* Treatment with systemic immunostimulatory agents or immunosuppressive medication
* Inadequately controlled arterial hypertension
* History of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease
* Evidence of bleeding diathesis or significant coagulopathy
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
* Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID)
* Preexisting renal impairment, myelosuppression, or hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (49):
- United States (5):
  - City of Hope Cancer Center, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke Cancer Center, Durham, North Carolina
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
- China (3):
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Zhongshan Hospital Fudan University, Shanghai
- Hong Kong (2):
  - Queen Mary Hospital; Dept. Of Haematology & Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Italy (4):
  - Fondazione Pascale; U.O. Sperimentazioni Cliniche, Napoli, Campania
  - Azienda Ospedaliero Universitaria di Bologna; Istituto di Ematologia "Lorenzo e Ariosto Seragnoli", Bologna, Emilia-Romagna
  - Istituto Clinico Humanitas - Humanitas Cancer Center, Rozzano, Sicily
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto
- Poland (5):
  - SP ZOZ Wojewódzki Szpital Specjalistyczny nr 4; Oddzial Onkologii Klinicznej, Bytom
  - Uniwersyteckie Centrum Kliniczne; Klinika Onkologii i Radioterapii, Gdansk
  - Szpital Wojewódzki im. Miko?aja Kopernika; Oddzia? Dzienny Chemioterapii, Koszalin
  - NIO im Marii Sklodowskiej-Curie; Klinika Onkologii i Radioterapii, Warsaw
  - Dolno?l?skie Centrum Onkologii; Oddzia? Onkologii Klinicznej i Chemioterapii, Wroc?aw
- Russia (4):
  - FSBI "National Medical Research Center of Oncology N.N. Blokhin?, Moscow, Moscow Oblast
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow, Moscow Oblast
  - SBIH "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of DHM", Moskva, Moscow Oblast
  - GBUZ Saint Petersburg Clinical Research Center of Specialized Types of Care (Oncology), Saint Petersburg, Sankt-Peterburg
- South Korea (5):
  - CHA Bundang Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Complejo Hospitalario de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron; Oncology, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Complejo Hospitalario de Orense; Servicio de Oncologia, Ourense
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Taiwan (2):
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Taipei Veterans General Hospital; Department of Oncology, Taipei
- Thailand (3):
  - Maharaj Nakorn Chiang Mai Hosp; Oncology Unit, Chiang Mai
  - Srinagarind Hospital; Medical Oncology Unit, Khon Kaen
  - Sunpasitthiprasong Hospital; Oncology and/or Hematology, Ubon Ratchathani
- Turkey (Türkiye) (4):
  - Adana Ac?badem Hospital Oncology Department, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
  - Koc Universitesi Hastanesi; T?bbi Onkoloji, Zeyt?nburnu
- Ukraine (3):
  - SI Institute of general&urgent surgery n/a Zaytseva V.T NAMSU, Kharkiv, Kharkiv Governorate
  - ?Kharkov Regional Oncology Center, Kharkiv, Kharkiv Governorate
  - SI "Shalimov National Institute of Surgery and Transplantation" of Nat.Acad of Med.Sci of Ukraine, Kyiv, KIEV Governorate
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital, London
  - Churchill Hospital, Oxford
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here ( https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Macarulla T, Ren Z, Chon HJ, Park JO, Kim JW, Pressiani T, Li D, Zhukova L, Zhu AX, Chen MH, Hack SP, Wu S, Liu B, Guan X, Lu S, Wang Y, El-Khoueiry AB. Atezolizumab Plus Chemotherapy With or Without Bevacizumab in Advanced Biliary Tract Cancer: Clinical and Biomarker Data From the Randomized Phase II IMbrave151 Trial. J Clin Oncol. 2025 Feb 10;43(5):545-557. doi: 10.1200/JCO.24.00337. Epub 2024 Oct 18. PMID 39423355
- [Derived] Hack SP, Verret W, Mulla S, Liu B, Wang Y, Macarulla T, Ren Z, El-Khoueiry AB, Zhu AX. IMbrave 151: a randomized phase II trial of atezolizumab combined with bevacizumab and chemotherapy in patients with advanced biliary tract cancer. Ther Adv Med Oncol. 2021 Jul 31;13:17588359211036544. doi: 10.1177/17588359211036544. eCollection 2021. PMID 34377158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is considered "Completed" because all pre-planned study activities and analyses have been performed. Participants are ongoing treatment on a roll over study.
Groups:
- Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond); Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond): *Cycle is 21 days. Cisplatin is administered on Days 1 and 8 of each 21 day cycle for cycles 1-8.
Period: Overall Study
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Started | 83 | 79
Completed | 0 | 0
Not Completed | 83 | 79
Not completed — Death | 51 | 49
Not completed — Progressive Disease | 1 | 0
Not completed — Symptomatic Deterioration | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Study Terminated By Sponsor | 28 | 24
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond) | Total
Number analyzed (Participants) | 83 | 79 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (9.8) | 59.6 (9.9) | 61.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 30 | 75
  Male | 38 | 49 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 82 | 78 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 37 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 46 | 41 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first)
Time Frame: Randomization to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first)(up to approximately 14 months)
Population: Analysis was performed on the Intent-to-treat (ITT) population, defined as all randomized participants, regardless of whether they received the assigned treatment or not, were included for analyses with participants grouped according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Number analyzed (Participants) | 83 | 79
Months | 7.92 [6.18 to 8.41] | 8.35 [6.83 to 9.96]
Statistical Analysis 1: Comparison: Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) vs Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond); Stratified analysis. Stratification factors are: Location of primary tumor (iCCA vs. eCCA vs. GBC), Geographic region (Asia vs. Rest of the World); Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.51 to 1.14]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: Randomization to death from any cause (up to approximately 23 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Number analyzed (Participants) | 83 | 79
Months | 14.59 [11.17 to NA] — With ~60% events to patients ratio, this happens due to no events occurred at the timepoint in the upper end required per the non-parameteric estimation method of Brookmeyer-Crowley. | 14.85 [11.63 to 17.97]
Statistical Analysis 1: Comparison: Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) vs Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8857, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.64 to 1.47]

3. Secondary Outcome: Confirmed Objective Response Rate (ORR)
Description: Confirmed ORR is defined as the proportion of participants with Complete Response (CR) or Partial Response (PR) on two consecutive occasions >=4 weeks apart, as determined by the investigator according to RECIST v1.1.
Time Frame: Randomization up to approximately 14 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Number analyzed (Participants) | 83 | 79
Percentage of participants | 25.3 | 24.1

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first occurrence of a confirmed objective response to disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first).
Time Frame: First occurrence of a confirmed objective response to disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first)(up to approximately 14 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Number analyzed (Participants) | 21 | 19
Months | 5.78 [4.27 to 6.70] | NA [6.44 to NA] — Insufficient number of participants with events.

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the proportion of participants with a CR or a PR on two consecutive occasions >= 4 weeks apart or SD with a minimum duration of 9weeks, as determined by the investigator according to RECIST v1.1
Time Frame: Randomization up to approximately 14 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Number analyzed (Participants) | 83 | 79
Percentage of participants | 75.9 | 78.5

6. Secondary Outcome: Time to Confirmed Deterioration (TTCD)
Description: TTCD in patient-reported physical functioning, role functioning, and quality of life, as measured by the respective scales of the EORTC QLQ-C30 and/or EORTC IL77, and defined as the time from randomization to the first clinically meaningful deterioration that is either maintained for two consecutive assessments or followed by death from any cause within 3 weeks.
Time Frame: Randomization to the first clinically meaningful deterioration (up to approximately 14 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Number analyzed (Participants) | 83 | 79
Months
  Quality of Life | 6.28 [3.06 to NA] — Insufficient number of participants with events. | 2.79 [1.58 to 5.32]
  Physical Function Scale | 3.29 [1.87 to 10.58] | 6.21 [4.63 to NA] — Insufficient number of participants with events.
  Role Function Scale | 3.52 [2.20 to 8.51] | 4.24 [2.10 to 6.28]
Statistical Analysis 1: Comparison: Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) vs Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond); Quality of Life; Test type: Superiority — Stratified analysis. Stratification factors are: Location of primary tumor (iCCA vs. eCCA vs. GBC), Geographic region (Asia vs. Rest of the World); Regression, Cox; Hazard Ratio (HR) = 1.56, 95% CI 2-sided [0.93 to 2.63]
Statistical Analysis 2: Comparison: Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) vs Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond); Physical Function Scale; Test type: Superiority — [test comment as in outcome 6, analysis 1]; Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.48 to 1.36]
Statistical Analysis 3: Comparison: Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) vs Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond); Role Function Scale; Test type: Superiority — [test comment as in outcome 6, analysis 1]; Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.68 to 1.85]

7. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: Percentage of participants with at least one adverse event.
Time Frame: Treatment start up to approximately 30 months.
Population: Safety analyses will be performed on the safety-evaluable population, which is defined as all randomized participants who receive any amount of any component of protocol treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
Number analyzed (Participants) | 81 | 78
Percentage of participants | 100 | 100

8. Secondary Outcome: Serum Concentration of Atezolizumab
Description: Serum concentration of atezolizumab at specified timepoints.
Time Frame: Pre-Dose on Day 1 of Cycles 1, 2, 3, 4, 8, 12, and 16, and Post Dose Day 1 of Cycle 1 (cycle length=21 days)
Population: The PK analysis population consisted of all participants with at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: μg/ mL
Arm/Group | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond) | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond)
Number analyzed (Participants) | 78 | 81
μg/ mL
  Cycle 1 Day 1 Pre-Dose: number analyzed (Participants) | 74 | 78
  Cycle 1 Day 1 Pre-Dose | NA (NA) — Below the level of detection. | NA (NA) — Below the level of detection.
  Cycle 1 Day 1 Post Dose: number analyzed (Participants) | 78 | 80
  Cycle 1 Day 1 Post Dose | 411 (73.8) | 416 (173)
  Cycle 2 Day 1 Pre-Dose: number analyzed (Participants) | 75 | 78
  Cycle 2 Day 1 Pre-Dose | 79.4 (46.1) | 85.0 (71.7)
  Cycle 3 Day 1 Pre-Dose: number analyzed (Participants) | 72 | 74
  Cycle 3 Day 1 Pre-Dose | 118 (41.4) | 129 (83.5)
  Cycle 4 Day 1 Pre-Dose: number analyzed (Participants) | 69 | 64
  Cycle 4 Day 1 Pre-Dose | 155 (50.6) | 153 (74.8)
  Cycle 8 Day 1 Pre-Dose: number analyzed (Participants) | 54 | 51
  Cycle 8 Day 1 Pre-Dose | 200 (100) | 224 (126)
  Cycle 12 Day 1 Pre-Dose: number analyzed (Participants) | 31 | 28
  Cycle 12 Day 1 Pre-Dose | 210 (76.4) | 223 (103)
  Cycle 16 Day 1 Pre-Dose: number analyzed (Participants) | 8 | 6
  Cycle 16 Day 1 Pre-Dose | 174 (64.9) | 230 (71.6)

9. Secondary Outcome: Prevalence of ADAs to Atezolizumab
Time Frame: Baseline
Population: The immunogenicity analysis population consist of all participants with at least 1 postbaseline ADA assessment. Participants are grouped according to treatment received. No data were collected because the study was discontinued before any measurements were completed.
Arm/Group | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond) | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence of ADAs to Atezolizumab
Time Frame: At pre-defined intervals from administration of study drug up to approximately 14 months
Population: as for outcome 9
Arm/Group | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond) | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first study drug until the data cut-off on 25 August 2023 (up to approximately 30 months)
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. Serious & other adverse events reported based on safety population, which included participants who received any amount of any study drug.
Arm/Group | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond)
All-Cause Mortality (participants affected / at risk) | 51/83 | 49/79
Serious Adverse Events (participants affected / at risk) | 43/81 | 36/78
Other Adverse Events (participants affected / at risk) | 81/81 | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) (N=81) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond) (N=78)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (10) | 3 (5)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 5 (5) | 2 (3)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Recurrent pyogenic cholangitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Ocular myasthenia (Eye disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (2) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haematological infection (Infections and infestations) | 1 (2) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B: Atezo+PBO+CisGem (Cycle*1-8), Followed by Atezo+PBO (Cycle*9 and Beyond) (N=81) | Arm A: Atezo+Bev+CisGem (Cycle*1-8), Followed by Atezo+Bev (Cycle*9 and Beyond) (N=78)
Anaemia (Blood and lymphatic system disorders) | 51 (88) | 37 (59)
Neutropenia (Blood and lymphatic system disorders) | 17 (31) | 17 (37)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (13) | 7 (18)
Hypothyroidism (Endocrine disorders) | 6 (6) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 13 (16) | 15 (16)
Ascites (Gastrointestinal disorders) | 5 (5) | 5 (6)
Constipation (Gastrointestinal disorders) | 23 (25) | 30 (39)
Diarrhoea (Gastrointestinal disorders) | 13 (16) | 14 (22)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 32 (44) | 32 (51)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 10 (10)
Vomiting (Gastrointestinal disorders) | 12 (12) | 16 (23)
Asthenia (General disorders) | 16 (33) | 14 (28)
Fatigue (General disorders) | 18 (22) | 21 (29)
Oedema peripheral (General disorders) | 7 (8) | 6 (6)
Pyrexia (General disorders) | 20 (44) | 14 (26)
COVID-19 (Infections and infestations) | 13 (13) | 11 (12)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (4)
Alanine aminotransferase increased (Investigations) | 15 (22) | 11 (15)
Aspartate aminotransferase increased (Investigations) | 17 (20) | 10 (15)
Blood alkaline phosphatase increased (Investigations) | 5 (7) | 5 (9)
Blood bilirubin increased (Investigations) | 7 (11) | 8 (8)
Blood creatinine increased (Investigations) | 11 (13) | 7 (7)
Lymphocyte count decreased (Investigations) | 7 (19) | 7 (17)
Neutrophil count decreased (Investigations) | 32 (80) | 38 (93)
Platelet count decreased (Investigations) | 22 (49) | 22 (48)
Weight decreased (Investigations) | 7 (7) | 10 (10)
Weight increased (Investigations) | 5 (5) | 5 (5)
White blood cell count decreased (Investigations) | 13 (34) | 15 (32)
Decreased appetite (Metabolism and nutrition disorders) | 14 (15) | 15 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (6) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (14) | 6 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (12) | 10 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (12) | 7 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (13)
Dizziness (Nervous system disorders) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 5 (8) | 7 (7)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (3)
Proteinuria (Renal and urinary disorders) | 9 (9) | 16 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 11 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (11) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 11 (15)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Hypertension (Vascular disorders) | 15 (17) | 29 (36)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 4 (4)
Mucosal inflammation (General disorders) | 2 (3) | 4 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT04677504/Prot_SAP_000.pdf